CLINICAL TRIAL: NCT07355231
Title: Lung Functional Avoidance Radiotherapy Using Hyperpolarized Xenon MRI
Acronym: GuidedRT
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xemed LLC (Industry)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MagniXene-255434
Record Dates: First submitted 2026-01-19; First posted 2026-01-21 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: lung cancer; non-small-cell lung cancer; radiation therapy; guided radiation therapy; functional lung avoidance; hyperpolarized xenon; HXe MRI
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Phase 1: open trial for establishing safety and methodology.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Guided Radiation Therapy for lung cancer using HXe MRI for functional lung avoidance and diagnosis. (Experimental): Patients with non-small cell lung cancer scheduled for radiation therapy will be voluntarily enrolled in this study. They will have their lung ventilation and function imaged with hyperpolarized xenon MRI. The 3D HXe images will be used in determining a functional lung avoidance treatment map. Patients will follow radiation therapy optimized for functional lung avoidance. At 6-month follow up the subjects will be imaged again with HXe to assess lung ventilation and function post-RT compared to baseline (pre-RT). Additionally, standard-of-care lung testing (DLCO, PFT) and quality-of-life questionnaires will be assessed at several time points during the study.
  Interventions: Combination Product: Hyperpolarized xenon MRI

INTERVENTIONS:
Combination Product: Hyperpolarized xenon MRI — Patients with non-small cell lung cancer scheduled for radiation therapy willing to take part in this study will undergo hyperpolarized xenon MRI at several time points prior and post RT. Images will be used to determine radiation treatment maps for functional lung avoidance. Reported adverse events caused by radiation induced lung injury and post-RT changes in the lung function will be compared to standard-of-care.

SUMMARY:
Cancer radiation treatment plans that employ lung functional avoidance methods require 3D maps that differentiate regions of healthy lung function from regions of functional compromised tissue to deliver sufficient dose to the tumor while preserving as much functioning lung as possible. Hyperpolarized xenon-129 MRI can provide maps of ventilatory function and gas exchange to the bloodstream. Improving treatment plans based on this novel imaging modality could reduce risk or severity of radiation pneumonitis and improve post-treatment quality of life.

DETAILED DESCRIPTION:
Customized 3D planning of radiation therapy for lung cancer delivers a lethal dose to the tumor region while avoiding important structures (spine) and organs (esophagus, heart, lungs). Since radiation dose to functioning lung is associated with acute radiation pneumonitis and chronic radiation fibrosis, researchers seek to shift dosage preferentially away from lung regions with highest function. Several lung functional imaging modalities have been investigated (ventilation-perfusion SPECT and PET, 4DCT, hyperpolarized 3He). These studies indicate that regional ventilation is not the optimal biometric. What is needed is a high-resolution imaging modality, tolerable to patients who have difficulty holding their breath, that delineates regions of full lung function warranting preservation, and also identifies regions whose function is irrevocably gone.

The investigators propose a translational study applying Hyperpolarized Xenon (HXe) MRI to improve lung-health outcomes for lung cancer patients treated with radiation therapy. This study will focus on a patient cohort with significant heterogeneity: new patients with lung cancer and GOLD stage 3+ emphysema as a comorbidity and patients receiving RT for their second (primary) lung cancer. Optimizing radiation therapy treatment plans could provide a statistically significant benefit within a manageably small patient cohort. Maps will delineate three regions of functionality: regions of full function, having both ventilation and gas exchange to blood (where radiation should be avoided or minimized), regions where function is irrevocably absent (where radiation dose can be increased/maximized), and regions where function may be present or recoverable (where radiation should remain below or at the normal dose limit). Regions of lungs with absent function will have highest priority for receiving radiation during the RT procedure, while healthy regions will be avoided. It is expected that following this functional avoidance procedure will result in a decrease in the radiation induced lung injury reported events and a better outcome of the radiation treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years with a diagnosis of non-small lung cancer and planned for a definitive course of radiation therapy.
* Preferred patients will have had successful radiation therapy for a prior lung cancer and developed a secondary lung cancer for which are to be treated.
* Other de-nuovo lung cancer patients planned for radiation therapy with lung heterogeneity from natural co-morbidities (e.g., COPD stage 3+).

Exclusion Criteria:

* Patients less than 18 years old
* Patients known to be pregnant - a positive pregnancy test will be used to respectively exclude pregnant patients,
* Any known contraindication to MRI examination
* Anyone with an implanted metal device
* Inability to provide informed consent
* A language, communication, cognitive or behavioral impairment that might interfere with fully informed participation in the study.
* History of uncompensated organ failure (i.e. organ failure that is not stabilized through medical intervention), which will be assessed by the PI.
* Homelessness or other unstable living situation
* Active drug or alcohol dependence
* Claustrophobia
* Subjects weighting more than 300 pounds.
* Subjects with chest size larger than the bore of MRI machine can accommodate

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-02-29 (Estimated); Study Completion 2028-02-29 (Estimated)

PRIMARY OUTCOMES:
Changes in DLCO at 6-month post RT treatment. | 1-year
  Subjects will have measurements of DLCO at baseline (before RT) and at 6-month post RT. An independent-sample t-test will be used to compare change in DLCO.

SECONDARY OUTCOMES:
Change in Quality of Life questionnaires from baseline to 6-month post-RT. | 1-year
  Quality of Life questionnaires ("MD Anderson Symptom Inventory - Lung Cancer" and "UCSD Shortness of Breath Questionnaire") will be assessed at baseline (prior to RT) and 6-month post RT. A independent-sample t-test will be used to compare changes in the QoL.
Change in HXe lung MRI metrics from baseline to 6-month post-RT. | 1-year
  HXe MRI metrics (including dynamic ventilation and dissolved phase - S/V and q-dot) will be assessed at baseline (prior to RT) and 6-month post RT. A independent-sample t-test will be used to compare changes in the HXe metrics.
Change in FEV1 from baseline to 6-month post-RT. | 1-year
  Other spirometry measurements (besides DLCO) such as FEV1, will be assessed at baseline (prior to RT) and 6-month post RT. A independent-sample t-test will be used to compare changes in FEV1.
Incidence/severity of pneumonitis. | 1-year
  Incidence/severity of pneumonitis will be graded using CTCAE at 6-month post RT. This will be compared with known results from standard-of-care RT.

IPD SHARING:
Plan to Share IPD: No